CLINICAL TRIAL: NCT05621343
Title: New Strategies for Assessment of the Persistence of Viable Bacilli in Latent and Active Tuberculosis
Acronym: TB-LIVE
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-04885
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-04

CONDITIONS: Latent Tuberculosis; Persistent Infection; Mycobacterium Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis; Persistent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Latent TB on treatment: Treatment according to existing Swedish guidelines with:
  Oral rifampicin 10 mg/kg (max 600mg) once daily during 4 months OR Oral isoniazide 5 mg/kg (max 300mg) once daily in combination with 40mg vitamin B6 (pyridoxin) during 6 months
- Latent TB not on treatment: Latent TB without indication for treatment OR patient who do not want to receive treatment
- Active TB with treatment: Treatment according to existing Swedish guidelines. Duration and choice of antibiotic therapy depending on the condition.
- Healthy control: Healthy

SUMMARY:
Current diagnostic tools such as interferon gamma release assay (IGRA) and purified protein derivative (PPD) can not distinguish patients with latent tuberculosis infection (LTBI) and persistence of live mycobacteria. This inability to rule out living mycobacteria in patients investigated for LTBI leads to unnecessary and potentially harmful treatment regimes all around the globe.

The goal of this observational study is to identify candidate biomarkers for viable bacilli in latent tuberculosis in order to decrease the use of unnecessary and ineffective antibiotic treatment.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the second leading cause of death due to a single infectious agent, with the main burden in resource-limited settings and in vulnerable populations. It is estimated that approximately 25% of the global population is infected with TB. LTBI is a condition where the mycobacteria rests within the body instead of creating active disease. About half of the active TB cases develop within 2 years of exposure and the other half reactivates as distant as several decades post exposure. Persistence of viable bacilli is a prerequisite for the reactivation of TB.

Through sampling of peripheral blood the investigators will investigate how selected cytokines, enzyme activity and gene expression changes during course of treatment, 4-6 months, and during follow up, 1 year. These patterns will be compared to the patterns of patients with: latent TB without treatment, active TB with treatment as well as healthy controls. Samples will be drawn at 0, 1, 6 and 12 months, after treatment initialization when applicable. Healthy controls will only be sampled once. Most of the analysis will be performed on TB-antigen stimulated blood.

The investigators hypothesize that there is a substantial fraction of latent TB patients who do not harbor live mycobacteria and that this is reflected in study outcome measures when given treatment. Furthermore, the investigators hypothesize that this fraction of latent TB patients will resemble healthy controls in terms of outcome measures whereas their counterpart, latent TB patients harboring living bacteria, will not.

ELIGIBILITY:
LTBI (2 groups)

Inclusion Criteria:

* latent tuberculosis: Interferon gamma (IFN-γ) >0.70 IU/ml in the Quantiferon-TB Plus assay
* age 15-25 years OR high likelihood of recent TB transmission
* informed consent

Exclusion Criteria:

* active tuberculosis
* chronic illness
* immunosuppressive treatment
* pregnancy (including 6 months post-partum)
* previous treatment for either active or latent TB infection

Controls

Inclusion Criteria:

* age 15-25 years
* informed consent

Exclusion Criteria:

* latent- OR active tuberculosis
* chronic illness
* immunosuppressive treatment
* pregnancy (including 6 months post-partum)
* previous treatment for either active or latent TB infection

Active TB

Inclusion Criteria:

* diagnosed with active TB
* informed consent

Exclusion Criteria:

age < 15 years

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals 15 years or older diagnosed with latent- or active tuberculosis or found healthy as part of routine care at the out- and inpatient department of the department for infectious diseases at Skåne University Hospital in Malmö, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cytokine levels | 0-12 months
  To determine levels of selected cytokines in supernatants of Mtb-incubated whole blood obtained from persons diagnosed with LTBI during the course of treatment, and to identify patterns of cytokine expression suggestive of bacterial eradication.
Gene expression | 0-12 months
  To characterize patterns of small non-coding RNA (sncRNA) expression (including microRNAs) in blood and plasma from persons diagnosed with LTBI, and to identify patterns of sncRNA expression in individuals with LTBI suggestive of bacterial eradication.
Activity of indoleamine 2, 3-dioxygenase (IDO) | 0-12 months
  3. To characterize IDO activity in plasma from persons diagnosed with LTBI, and to determine whether changes in IDO activity during the course of LTBI reflect bacterial eradication

CONTACTS AND LOCATIONS:
Overall Officials: Per Björkman, Professor, Principal Investigator — Lund University, Faculty of Medicine, Department of Translational Medicine
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Holmberg P, Janouskova M, Schmidt T, Neumann A, Olsson O, Isberg PE, Reimann M, Riesbeck K, Skogmar S, Bjorkman P. Blood levels of Mycobacterium tuberculosis (Mtb)antigen-triggered immune markers in people exposed to tuberculosis with regard to Mtb infection status and receipt of tuberculosis preventive therapy. Tuberculosis (Edinb). 2025 Mar;151:102595. doi: 10.1016/j.tube.2024.102595. Epub 2024 Dec 20. PMID 39742565